CLINICAL TRIAL: NCT06642272
Title: A Pragmatic Trial Comparing Empagliflozin and Dapagliflozin Through Cluster Randomization Embedded in the Electronic Health Record
Acronym: APPLE TREE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Daniel Mølager Christensen, Investigator, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2401312
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus, Type 2; Heart Failure; Chronic Kidney Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Failure; Renal Insufficiency, Chronic | interventions — empagliflozin; dapagliflozin

STUDY DESIGN:
Masking Description: Treatment assignment will be blinded to the statistician analysing the trial data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin 10 MG (Other): Head-to-head comparator
  Interventions: Drug: Empagliflozin 10 MG
- Dapagliflozin 10 MG (Other): Head-to-head comparator
  Interventions: Drug: Dapagliflozin 10 MG

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Once daily
  Arms: Empagliflozin 10 MG
Drug: Dapagliflozin 10 MG — Once daily
  Arms: Dapagliflozin 10 MG

SUMMARY:
The aim of this clinical trial is investigate the comparative effectiveness of empagliflozin and dapagliflozin for the treatment of diabetes, chronic kidney disease, and heart failure.

Patients who are prescribed either empagliflozin or dapagliflozin, as part of daily clinical practice at the participating sites, will be included in the study. Treatment will be randomized automatically through the electronic health record software in clusters defined by time of day.

https://www.appletreestudy.com

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or more

Exclusion Criteria:

* Incapabability of giving informed consent
* Withdrawal of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17200 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to the first occurrence of any of the components of the composite: all-cause mortality, hospitalization for heart failure, hospitalization for myocardial infarction, hospitalization for ischemic stroke, and incident or worsening nephropathy. | Up to 24 months
  Incident or worsening nephropathy is defined as:
  * A sustained decrease in estimated glomerular filtration rate (eGFR) of ≥40% from baseline
  * A sustained decrease in eGFR of ≤10 per minute per 1.73 m2
  * Initiation of dialysis
  * Kidney transplantation

SECONDARY OUTCOMES:
All-cause mortality | Up to 24 months
Hospitalization for heart failure | Up to 24 months
Hospitalization for myocardial infarction | Up to 24 months
Hospitalization for ischemic stroke | Up to 24 months
Incident or worsening nephropathy | Up to 24 months
  Defined as a sustained decrease in estimated glomerular filtration rate (eGFR) of ≥40% from baseline, a sustained decrease in eGFR of ≤10 per minute per 1.73 m2, initiation of dialysis, or kidney transplantation
Hospitalization for coronary revascularization | Up to 24 months
Hospitalization for unstable angina | Up to 24 months

OTHER OUTCOMES:
Hospitalization for ketoacidosis | Up to 24 months
  Safety outcome
Hospitalization for limb amputation | Up to 24 months
  Safety outcome
Hospitalization for genitourinary infection | Up to 24 months
  Safety outcome
Hospitalization for fracture | Up to 24 months
  Safety outcome

CONTACTS AND LOCATIONS:
Locations (12):
- Denmark (12):
  - Bispebjerg Hospital, Copenhagen
  - Rigshospitalet, Copenhagen
  - Herlev and Gentofte Hospital, Herlev
  - Steno Diabetes Center Copenhagen, Herlev
  - Nordsjællands Hospital, Hillerød
  - Holbæk Sygehus, Holbæk
  - Hvidovre Hospital, Hvidovre
  - Sjællands Universitetshospital, Køge
  - Nykøbing F. Sygehus, Nykøbing Falster
  - Sjællands Universitetshospital, Roskilde
  - Bornholms Hospital, Rønne
  - Slagelse Sygehus, Slagelse